CLINICAL TRIAL: NCT06266897
Title: A Study on the Correlation Between Endometriosis and Intra-tissue Microbiota
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZhujiangEM
Record Dates: First submitted 2024-01-25; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Endometriosis
Keywords: Microbiota; Microbiome; Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We will obtain serum, vaginal swabs, cervical mucus, and feces from the participant before surgery. We will also collect peritoneal fluid, eutopic endometrium, and ectopic endometrium lesion if the surgical approach allows.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EM group: Patient diagnosed with endometriosis after confirmation by laparoscopic surgery and pathologic examination.
- Control group: Patient diagnosed without endometriosis after confirmation by laparoscopic surgery and pathologic examination, usually with benign gynecologic conditions such as uterine fibroids or teratomas.

SUMMARY:
Endometriosis (EM) is a common gynecological condition, but the pathogenesis of it has not yet been clarified. Here, the investigators wanted to investigate the correlation between endometriosis and the intra-tissue microbiota. The investigators planed to collect serum, vaginal swabs, cervical mucus, feces, peritoneal fluid, and endometrial tissue for sequencing and experiments.

DETAILED DESCRIPTION:
Endometriosis (EM) is a common gynecological condition that occurs in women of reproductive age and is characterized by pain, masses, and infertility. EM is a tumor-like disease that is invasive, metastatic, recurrent, but the pathogenesis of EM has not yet been clarified. Advances in the study of intratumoral microbiota provided increasing evidence confirming the presence and mechanism of bacteria in tumor tissues. Therefore, the investigators wanted to investigate the correlation between endometriosis and its microbiota in the endometrial tissue.

Participants in this study will be recruited in the obstetrics and Obstetrics and Gynecology Medical Center of Zhujiang Hospital. With reference to the inclusion and exclusion criteria, patients admitted for surgery were under screening. Participants were assigned to Endometriosis group after confirmation by laparoscopy together with biopsy analysis, while the control group was identified as non-EM patients, usually with benign gynecologic conditions such as uterine fibroids or teratomas.

The investigators will obtain serum, vaginal swabs, cervical mucus, and feces from the participant before surgery. The peritoneal fluid, eutopic endometrium, and ectopic endometrium lesion will also be collected if the surgical approach allows. The specimens will be sent for microbiota sequencing, transcriptome sequencing, metabolome sequencing, single cell sequencing, and laboratory experiments.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-52 years old.
2. Regular menstruation with a cycle of 28-35 days.
3. No sexual intercourse 1 week before the operation.
4. No systemic or local use of antibiotics and probiotics for 6 months prior to surgery.
5. No history of acute or chronic pelvic inflammatory disease.
6. Subjects fully understand the significance of the study and sign the informed consent form.

Exclusion Criteria:

1. In pregnancy.
2. Intraoperative conditions or pathological examination suggest a malignant or junctional disease.
3. Severe anatomical abnormalities of the pelvis.
4. Pelvic contamination with large amounts of blood during laparoscopic operation.
5. History of gene therapy, blood transfusion, stem cell therapy, or bone marrow transplantation
6. Psychiatric, personality disorders, or abuse of psychoactive substances.
7. Immunodeficiencies, allergies, or autoimmune diseases.
8. Contraindications to endotracheal intubation anesthesia.
9. Absolute or relative contraindications to laparoscopic or hysteroscopic surgery.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants in this study will be recruited in the obstetrics and Obstetrics and Gynecology Medical Center of Zhujiang Hospital. With reference to the inclusion and exclusion criteria, patients admitted for surgery were under screening.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Metagenomics Next Generation Sequencing of the Intra-tissue Microbiota Composition | 3 years
  Using metagenomics sequencing of microbiota, compare the microbial composition differences of specimens derived from EM group and control group, including the alpha diversity(Shannon index, Simpson index, etc.), beta diversity(PCoA analysis, Bray-Curtis, etc.) differential taxonomy, and KEGG pathway prediction.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Ma, PhD, Principal Investigator — Zhujiang Hospital, Southern Medical University, China
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China